CLINICAL TRIAL: NCT01263782
Title: BATTLE-FL: A Biomarker-Integrated Study in Patients With Advanced Non-Small Cell Lung Cancer Treated in the Front-Line (FL) Setting
Brief Title: BATTLE-FL: Front-Line Biomarker-Integrated Treatment Study in Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Eli Lilly and Company (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0097; NCI-2011-00301 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-12-17; First posted 2010-12-21 (Estimated); Results first posted 2019-05-08 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Lung Cancer
Keywords: Non-Small Cell Lung Cancer; NSCLL; Nonsquamous cell; Metastatic disease; Cixutumumab; IMC-A12; Carboplatin; Paraplatin; Pemetrexed; LY231514; Alimta; MTA; Multitargeted Antifolate; NSC-698037; Bevacizumab; Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — Carboplatin; Pemetrexed; Bevacizumab; cixutumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Carboplatin + Pemetrexed (Experimental): The chemotherapy will be Carboplatin (AUC 6) and Pemetrexed (500 mg/m2) every 3 weeks for 4 cycles.
  Then maintenance Pemetrexed (500 mg/m2 every 3 weeks) will be administered until disease progression or excessive toxicity.
  If patients are randomized into one of the arms with a biologic therapy, patients will take the chemotherapy prescribed above, but will also receive the biologic therapy during the same time period.
  Interventions: Drug: Carboplatin; Drug: Pemetrexed
- Chemo (Carbo/Peme) + Bevacizumab (Experimental): Carboplatin AUC 6 by vein on day 1 of every 21 day cycle for 4 cycles. Pemetrexed 500 mg/m2 by vein on day 1 of each 21 day cycle. Bevacizumab 15 mg/kg by vein on day 1 of each 21 day cycle.
  Interventions: Drug: Carboplatin; Drug: Pemetrexed; Drug: Bevacizumab
- Chemo (Carbo/Peme) (Experimental): Carboplatin AUC 6 by vein on day 1 of every 21 day cycle for 4 cycles. Pemetrexed 500 mg/m2 by vein on day 1 of each 21 day cycle.
  Interventions: Drug: Carboplatin; Drug: Pemetrexed
- Chemo (Carbo/Peme) + Cixutumumab (Experimental): Carboplatin AUC 6 by vein on day 1 of every 21 day cycle for 4 cycles. Pemetrexed 500 mg/m2 by vein on day 1 of each 21 day cycle.
  Cixutumumab 20 mg/kg by vein on day 1 of each 21 day cycle.
  Interventions: Drug: Carboplatin; Drug: Pemetrexed; Drug: Cixutumumab

INTERVENTIONS:
Drug: Carboplatin — AUC 6 by vein on day 1 of every 21 day cycle for 4 cycles.
  Other Names: Paraplatin
Drug: Pemetrexed — 500 mg/m2 by vein on day 1 of each 21 day cycle.
  Other Names: LY231514; Alimta; MTA; Multitargeted Antifolate; NSC-698037
Drug: Bevacizumab — 15 mg/kg by vein on day 1 of each 21 day cycle.
  Other Names: Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
  Arms: Chemo (Carbo/Peme) + Bevacizumab
Drug: Cixutumumab — 20 mg/kg by vein on day 1 of each 21 day cycle.
  Other Names: IMC-A12
  Arms: Chemo (Carbo/Peme) + Cixutumumab

SUMMARY:
The goal of this clinical research study is to learn if knowing biomarker status can help researchers find better treatment combinations for patients with advanced NSCLC.

Researchers want to use biomarker status to decide what drug (bevacizumab, or cixutumumab) to give in combination with carboplatin and pemetrexed. The safety of these drug combinations will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Carboplatin is designed to interfere with the growth of cancer cells by stopping cell division, which may cause the cells to die.

Pemetrexed is designed to block enzymes in the body that play a part in tumor growth.

Bevacizumab is designed to block the growth of blood vessels that supply nutrients necessary for tumor growth. This may prevent or slow down the growth of cancer cells.

Cixutumumab is a monoclonal antibody, which means that it attaches to specific targets on cancer cells. These targets are called IGF-1R and help the cancer cells grow and divide. Cixutumumab is designed to block these receptors on tumor cells that may cause tumors to grow.

Study Groups and Drug Administration (Combination Therapy):

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the roll of dice) to 1 of 3 groups. You will have an equal chance of being assigned to each group. Each cycle is 21 days (+/- 5 days).

* If you are in Group 1, you will receive carboplatin and pemetrexed on Day 1 of each cycle. Carboplatin will be given by vein over 10 minutes. Pemetrexed will be given by vein over 30 minutes.
* If you are in Group 2, you will receive bevacizumab, carboplatin, and pemetrexed on Day 1 of each cycle. Bevacizumab will be given by vein over about 90 minutes for the first dose, about 60 minutes for the second dose, and about 30 minutes for all other doses. Carboplatin will be given by vein over 10 minutes. Pemetrexed will be given by vein over 30 minutes.
* If you are in Group 3, you will receive cixutumumab, carboplatin, and pemetrexed on Day 1 of each cycle. Cixutumumab is given by vein over 60 minutes. Carboplatin will be given by vein over 10 minutes. Pemetrexed will be given by vein over 30 minutes.

Study Visits During Combination Therapy:

If you are in Group 3, before you begin receiving study drugs, you will have a hearing test.

On Day 1 (+/- 5 days) of Cycles 1, 2, and 4:

* You will have a physical exam, including measurement of your weight and vital signs.
* You will be asked about any drugs you may be taking and any side effects you may be having.
* Your performance status will be recorded.
* Blood (about 3 teaspoons) will be drawn for routine tests.
* If you are in Group 2, urine will be collected for routine tests.

On Days 8 and 15 of Cycle 1:

°If you are in Group 3, blood (about 1 teaspoon) will be drawn for routine tests.

On Day 1 of Cycle 3:

* You will have a physical exam, including measurement of your weight and vital signs.
* You will be asked about any drugs you may be taking and any side effects you may be having.
* Your performance status will be recorded.
* Blood (about 3 teaspoons) will be drawn for routine tests.
* You will have a CT scan and/or MRI scan of the chest (and abdomen if the doctor thinks it is needed) to check the status of the disease.
* You will have an MRI scan of the brain.
* You will have a chest x-ray to check the status of the disease.
* If you are in Group 2, urine will be collected for routine tests.

At any time your doctor thinks it may be needed, blood (about 1 teaspoon) will be drawn to check how well your blood clots.

Maintenance Therapy:

After you have completed 4 cycles of combination therapy, you may be eligible for maintenance therapy.

If you are in Group 1,you will receive pemetrexed by vein over 10 minutes on Day 1 (± 5 days) of every 21-day cycle.

If you are in Group 2, you will receive pemetrexed by vein over 10 minutes and bevacizumab over about 30 minutes on Day 1 (± 5 days) of every 21-day cycle.

If you are in Group 3, you will receive pemetrexed by vein over about 10 minutes and cixutumumab by vein over about 60 minutes on Day 1 (± 5 days) of every 21-day cycle.

Study Visits During Maintenance Therapy:

On Day 1 of each cycle:

* You will have a physical exam, including measurement of your weight and vital signs.
* You will be asked about any drugs you may be taking and any side effects you may be having.
* Your performance status will be recorded.
* Blood (about 3 teaspoons) will be drawn for routine tests.
* You will have a CT scan and/or MRI scan of the chest (and abdomen if the doctor thinks it is needed) to check the status of the disease.
* You will have an MRI scan of the brain.
* You will have a chest x-ray to check the status of the disease.
* If you are in Group 2, urine will be collected for routine tests.

Length of Study:

You may continue taking the study drug(s) for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse or intolerable side effects occur.

Your participation on the study will be over once you have completed the end-of-dosing visit and follow-up.

End-of-Dosing Visit:

When you go off study for any reason, you will have an end-of-dosing visit. The following tests and procedures will be performed:

* Your medical history will be recorded.
* You will have a complete physical exam, including measurement of your weight and vital signs.
* You will be asked about any drugs you may be taking and any side effects you may be having.
* Your performance status will be recorded.
* Blood (about 3 teaspoons) and urine will be collected for routine tests.
* You will have a CT scan and/or MRI of the chest (and abdomen if the doctor thinks it is needed) to check the status of the disease.
* You will have an MRI scan of the brain.
* You will have a chest x-ray.
* You will have an ECG.
* If you are in Group 3, you will have a hearing test.

Follow-Up:

You will have follow-up every 4 weeks after you are no longer taking the study drugs. You will be contacted at a clinic visit or by phone. You will be called every 3 months for up to 3 years and asked about any cancer treatments you may be receiving. This phone call should take about 10 minutes.

This is an investigational study. Carboplatin and pemetrexed are FDA approved and commercially available for the treatment of certain types of NSCLC. Bevacizumab is FDA approved and commercially available for treatment of certain types of colon or rectal cancer, NSCLC, and renal cell carcinoma. Cixutumumab is not FDA approved or commercially available. At this time, cixutumumab is only being used in research.

Up to 225 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has a diagnosis of pathologically confirmed nonsquamous (nonpredominant squamous) NSCLC by tumor biopsy and/or fine-needle aspiration. Mixed tumors will be categorized by the predominant cell type; if small cell elements are present, the patient is ineligible.
2. The patient has a diagnosis of either stage IIIB or stage IV NSCLC or has recurrent NSCLC and is not a candidate for curative treatment. Patients may not have had chemotherapy for the advanced setting.
3. The patient has measurable NSCLC.
4. The patient's Eastern Cooperative Oncology Group (ECOG) performance status is </=2 at study entry.
5. The patient should have tumor available for epidermal growth factor receptor (EGFR) mutations, ALK fusions and other molecular analyses. If there is no tissue then the patient has should have biopsy accessible tumor.
6. The patient has adequate hematologic function as defined by an absolute neutrophil count (ANC) >/= 1,500/mm^3, platelet count >/= 100,000/mm^3, white blood cell count (WBC) >/= 3,000/ mm^3, and hemoglobin >/= 9 g/dL.
7. The patient has adequate hepatic function as defined by a total bilirubin level </= 1.5 X the upper limit of normal (Serum bilirubin >/= 1.5x Upper Limit of Normal in the setting of known Gilbert's disease is allowed), and alkaline phosphatase, AST and ALT </= 2.5 X the upper limit of normal or </= 5.0 x ULN if liver metastases are present.
8. The patient has adequate renal function as defined as CrCl of at least 45ml/min.
9. If patient has brain metastasis, they must have been stable (treated and/or asymptomatic) and off steroids for at least 2 weeks.
10. The patient is >/= 18 years of age.
11. The patient has signed informed consent.
12. Pregnancy Test. Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation and for six (6) months after discontinuation of the study drugs. Childbearing potential will be defined as women who have had menses within the past 12 months, who have not had tubal ligation, hysterectomy or bilateral oophorectomy. Should a woman become pregnant or suspect that she is pregnant while participating in this study, she should inform her treating physician immediately. The patient, if a man, agrees to use effective contraception or abstinence for the duration of study participation and for six (6) months after discontinuation of the study drugs.
13. The ability to interrupt the use of NSAIDS two days before (5 days for long-acting NSAIDs), the day of, and 2 days following administration of Pemetrexed.

Exclusion Criteria:

1. The patient has received prior definitive therapy (chemotherapy, surgery, or radiotherapy) within 3 months of initiating study drug or within, 2 weeks of localized palliative radiotherapy. Patients treated with initial biologic therapy that progress are eligible (no drug within 4 weeks). Patients must have recovered from the acute toxic effects prior to Day 1 of Cycle 1 to grade </= 1 or baseline.
2. Patients may not have had prior chemotherapy for first line treatment for NSCLC Stage IIIB/IV. Patient with activating EGFR mutations could have been treated with an EGFR tyrosine kinase inhibitor. Similarly patient with ALK or ROS1 fusions could have had treatment with crizotinib or other ALK inhibitors. Patients may not have had prior biologic therapy with antibodies targeting VEGF,or insulin-like growth factor receptor (IGFR).
3. The patient has undergone prior thoracic or abdominal surgery within 30 days of study entry, excluding prior diagnostic biopsy.
4. The patient has a history of uncontrolled angina, arrhythmias, or congestive heart failure.
5. The patient has inadequately controlled hypertension (defined as systolic blood pressure > 140 and/or diastolic > 90 mm Hg on antihypertensive medications).
6. The patient has a history of stroke or transient ischemic attack within 6 months prior to Day 1 of Cycle 1.
7. The patient is unable or unwilling to take folic acid, vitamin B12 supplementation, or dexamethasone according to protocol.
8. The patient has neuropathy >/= grade 2.
9. The patient has a history of gastrointestinal fistula, perforation, or abscess, inflammatory bowel disease, or diverticulitis.
10. The patient is currently receiving ongoing treatment with full-dose warfarin or equivalent (that is, unfractionated and/or low molecular weight heparin).
11. The patient is pregnant.
12. The patient is breastfeeding.
13. Presence of significant third space fluid which cannot be controlled by drainage.
14. The patient's tumor harbors the EML4-ALK fusion gene.
15. Drug Specific Eligibility for Treatment Arms. Patients are excluded from the Bevacizumab arm if they have a history of hemoptysis (>/= ½ teaspoon of bright red blood per episode) within 3 months prior to randomization.
16. Drug Specific Eligibility for Treatment Arms. Patients are excluded from Bevacizumab arm if the Urine Protein Creatinine (UPC) ratio is not within the institutional normal limits.
17. Drug Specific Eligibility for Treatment Arms. Patients are excluded from the IMC-A12 containing arm if they have poorly controlled diabetes: HBA1C>8% or if the patient has abnormally elevated fasting serum glucose (defined >110% ULN).
18. Drug Specific Eligibility for Treatment Arms. Patients are excluded if they have known hypersensitivity to any of the drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-05-17 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Simon, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-four patients with non-small cell lung cancer were recruited from June 2011 to October 2013 at the University of Texas MD Anderson Cancer Center.
Pre-assignment Details: The patients had pre-treatment evaluations, which were used to determine the patients' study eligibility, within 4 weeks prior to initiating therapy. Out of 64 participants, 40 was screen failed.
Groups:
- Carboplatin + Pemetrexed x 4 Cycles Followed by Maintenance Pe: Four 21-day cycles of combination AUC 6 of carboplatin and 500 mg/m2 of pemetrexed; maintenance pemetrexed and pemetrexed every 21 days until disease progression
- Carboplatin + Pemetrexed + Bevacizumab Followed by Maintenance: Four 21-day cycles of combination AUC 6 of carboplatin, 500 mg/m2 of pemetrexed, and 15 mg/kg of bevacizumab; maintenance pemetrexed and bevacizumab every 21 days until disease progression
- Carboplatin + Pemetrexed + Cetuximab Followed by Maintenance P: Four 21-day cycles of combination AUC 6 of carboplatin, 500 mg/m2 of pemetrexed, and 250 mg/m2 of cetuximab (400mg/m2 on Cycle 1, Day 1 only); maintenance pemetrexed and cetuximab every 21 days until disease progression
- Carboplatin + Pemetrexed + Cixutumumab Followed by Maintenance: Four 21-day cycles of combination AUC 6 of carboplatin, 500 mg/m2 of pemetrexed, and 20 mg/kg of cixutumumab; maintenance pemetrexed and cixutumumab every 21 days until disease progression
Period: Overall Study
Arm/Group | Carboplatin + Pemetrexed x 4 Cycles Followed by Maintenance Pe | Carboplatin + Pemetrexed + Bevacizumab Followed by Maintenance | Carboplatin + Pemetrexed + Cetuximab Followed by Maintenance P | Carboplatin + Pemetrexed + Cixutumumab Followed by Maintenance
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 3 | 5
Not Completed | 0 | 0 | 3 | 1
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Progressive disease | 0 | 0 | 0 | 1
Not completed — Too early | 0 | 0 | 1 | 0
Not completed — Inevaluable | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carboplatin + Pemetrexed x 4 Cycles Followed by Maintenance Pe | Carboplatin + Pemetrexed + Bevacizumab Followed by Maintenance | Carboplatin + Pemetrexed + Cetuximab Followed by Maintenance P | Carboplatin + Pemetrexed + Cixutumumab Followed by Maintenance | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 3 | 2 | 11
  >=65 years | 3 | 3 | 3 | 4 | 13
Age, Continuous [Median (Full Range); unit: years] | 66 [54 to 71] | 65 [56 to 75] | 68 [58 to 84] | 68 [55 to 73] | 66 [54 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 3 | 0 | 7
  Male | 3 | 5 | 3 | 6 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 0 | 0 | 3
  Unknown or Not Reported | 5 | 4 | 6 | 6 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 1 | 3
  White | 5 | 5 | 5 | 4 | 19
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 24

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: It is defined as from treatment start to the time of progression or death, whichever occurred first, or to the time of last contact. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From treatment start to the time of progression or death, whichever occurred first, or to the time of last contact, assessed up to 5 years
Population: Patients who had treatment
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Carboplatin + Pemetrexed x 4 Cycles Followed by Maintenance Pe | Carboplatin + Pemetrexed + Bevacizumab Followed by Maintenance | Carboplatin + Pemetrexed + Cetuximab Followed by Maintenance P | Carboplatin + Pemetrexed + Cixutumumab Followed by Maintenance
Number analyzed (Participants) | 6 | 6 | 6 | 6
month | 5.2 [1.3 to 11.2] | 14.5 [1.5 to 53.7] | 20.6 [1.4 to 26.0] | 8 [3.2 to 22.09]

2. Secondary Outcome: Overall Response Rate
Description: Tumor response was assessed every two cycles of completed therapy. Responses will be based on a comparison to the pretreatment tumor evaluation. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: From treatment start to every two cycles of completed therapy.
Population: Patients who were evaluable for response
Measure: Count of Participants; unit: Participants
Arm/Group | Carboplatin + Pemetrexed x 4 Cycles Followed by Maintenance Pe | Carboplatin + Pemetrexed + Bevacizumab Followed by Maintenance | Carboplatin + Pemetrexed + Cetuximab Followed by Maintenance P | Carboplatin + Pemetrexed + Cixutumumab Followed by Maintenance
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  No change/Stable Disease | 5 | 3 | 2 | 3
  Partial Remission | 0 | 3 | 1 | 2
  Progressive Disease | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 3 years
Description: Patients who were evaluable for toxicity and grades 1-3 adverse events.
Arm/Group | Carboplatin + Pemetrexed x 4 Cycles Followed by Maintenance Pe | Carboplatin + Pemetrexed + Bevacizumab Followed by Maintenance | Carboplatin + Pemetrexed + Cetuximab Followed by Maintenance P | Carboplatin + Pemetrexed + Cixutumumab Followed by Maintenance
All-Cause Mortality (participants affected / at risk) | 1/6 | 0/6 | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 2/6 | 0/6 | 2/3 | 0/5
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 3/3 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin + Pemetrexed x 4 Cycles Followed by Maintenance Pe (N=6) | Carboplatin + Pemetrexed + Bevacizumab Followed by Maintenance (N=6) | Carboplatin + Pemetrexed + Cetuximab Followed by Maintenance P (N=3) | Carboplatin + Pemetrexed + Cixutumumab Followed by Maintenance (N=5)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Other, Endarterectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than .26% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin + Pemetrexed x 4 Cycles Followed by Maintenance Pe (N=6) | Carboplatin + Pemetrexed + Bevacizumab Followed by Maintenance (N=6) | Carboplatin + Pemetrexed + Cetuximab Followed by Maintenance P (N=3) | Carboplatin + Pemetrexed + Cixutumumab Followed by Maintenance (N=5)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abrasions to RUE. (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (2) | 0 (0) | 1 (2)
Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaphylaxis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 3 (8) | 3 (6) | 2 (6) | 4 (8)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (5)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Billary tract infection (cholendocholithiasis) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CAD (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid Stenosis, Rt. interval (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholesterol high (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 2 (2) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 2 (2) | 2 (4) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1) | 1 (3)
Diverticulosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 4 (4) | 2 (2) | 2 (2)
Edema (Brain-cerebral) (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema face (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 1 (2) | 2 (2) | 1 (3)
Edema trunk (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Elevated LDH (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Esophageal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (5) | 4 (4) | 3 (3) | 4 (5)
Fever (General disorders) | 3 (4) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Glucosuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hearning Loss (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemoglobin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (10) | 1 (3) | 1 (1) | 3 (7)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (3) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (5) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (6) | 2 (2) | 3 (12) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Increasse LDH (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Irritability, intermittent (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 4 (4) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (4) | 2 (3) | 1 (2) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 4 (4) | 1 (1) | 2 (2)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (2) | 3 (4) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 2 (6) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Renal hemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
swelling both hands (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
White blood cell decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-03-07): https://cdn.clinicaltrials.gov/large-docs/82/NCT01263782/Prot_SAP_000.pdf